CLINICAL TRIAL: NCT00570037
Title: Prevention of Influenza in Infants by Immunization of Their Contacts in the Household
Brief Title: Feasibility of Cocooning Immunization Strategy With Influenza Vaccine
Acronym: Piiitch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00004990; 1U01IP000074-01 (NIH)
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Results first posted 2011-02-01 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2011-01

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Children
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunization Program (Active Comparator): Intervention Hospital - Standing postpartum vaccine orders, influenza vaccine clinic on postpartum ward for household contacts, mailed vaccine reminders
  Interventions: Biological: Trivalent inactivated influenza vaccine
- No Immunization Program (No Intervention): Comparison Hospital - Receipt of vaccine through routine clinical care

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Intramuscular injection, 0.5 mL or 0.25 mL depending on age of vaccine recipient, one or two doses administered a month apart depending on age and prior influenza vaccination history of recipient
  Other Names: Fluzone
  Arms: Immunization Program

SUMMARY:
Influenza causes epidemics of respiratory infection in young children each winter. Young children, particularly those under 6 months of age are most vulnerable to suffering from complications secondary to influenza infection. Consequently, influenza vaccine has been recommended for children 6-59 months of age. Influenza vaccine is not approved for use in children under 6 month of age who are at highest risk. Therefore, the Centers for Disease Control and Prevention Advisory Committee on Immunization Practices has recommended vaccination of household contacts of children under 6 month of age - a cocooning strategy.

The current study is a hospital-based study to assess the effectiveness of a program to vaccinate birth mothers and household contacts of newborns with influenza vaccine. We propose to study both birth mothers and household contacts of newborns delivered at Durham Regional Hospital and Duke University Medical Center, birthing hospitals serving Durham and surrounding counties in central North Carolina. We will implement several strategies to increase vaccine coverage rates at Durham Regional Hospital utilizing Duke University Hospital as a comparison setting. Strategies will include: standing vaccine orders for birth mothers, vaccine reminders for household contacts, and a hospital based influenza vaccine clinic to increase vaccine accessibility for household contacts. Vaccine coverage rates will be assessed utilizing a survey method (maternal interview at the birthing hospital and a follow-up telephone contact 6-8 weeks later). We hypothesize that influenza vaccine coverage rates for new mothers and household contacts of newborns delivered at the intervention hospital will be higher when compared to coverage rates in the comparison hospital. Demographic determinants of vaccine coverage and reasons for refusal of influenza vaccine will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Mother of a newborn delivered at either Durham Regional Hospital or Duke University Hospital between October 2007 and February 2008

Exclusion Criteria:

* Fetal demise or stillbirth
* Maternal rights relinquished
* Language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel B Walter, MD, MPH, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 2007 through February 2008 Post partum units of two Durham, North Carolina hospitals
Period: Overall Study
Arm/Group | Hospital With Immunization Program | Hospital With No Immunization Program
Started | 238 | 306
Completed | 194 | 237
Not Completed | 44 | 69
Not completed — Could not reach for 6-8 week contact | 44 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hospital With Immunization Program | Hospital With No Immunization Program | Total
Number analyzed (Participants) | 238 | 306 | 544
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 238 | 306 | 544
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 306 | 544
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 238 | 306 | 544

OUTCOME MEASURES:

1. Primary Outcome: Influenza Vaccine Coverage (Percent) for New Mothers of Newborns
Description: The percent of new mothers delivering at the hospital who reported receiving an influenza vaccine during their pregnancy, in the hospital after delivery, or during the 6 to 8 week postpartum period
Time Frame: Pregnancy period through 6 to 8 weeks postpartum
Measure: Number; unit: Percentage of Participants
Arm/Group | Hospital With Immunization Program | Hospital With No Immunization Program
Number analyzed (Participants) | 238 | 306
Percentage of Participants | 70 | 64

2. Primary Outcome: Influenza Vaccine Coverage (Percent) for New Fathers of Newborns
Description: The percent of new fathers who as reported by new mothers received an influenza vaccine during the mothers pregnancy, in the hospital after delivery, or during the 6 to 8 week period following the birth of their baby
Time Frame: Pregnancy period through 6 to 8 weeks postpartum
Measure: Number; unit: Percentage of Fathers of Newborns
Arm/Group | Hospital With Immunization Program | Hospital With No Immunization Program
Number analyzed (Participants) | 238 | 306
Percentage of Fathers of Newborns | 53 | 26

3. Primary Outcome: Influenza Vaccine Coverage (Percent) for All Household Contacts of Newborns
Description: The percent of all household contacts of newborns who as reported by new mothers received an influenza vaccine during the mothers pregnancy, in the hospital after delivery, or during the 6 to 8 week period following the birth of their baby
Time Frame: Pregnancy period through 6 to 8 weeks postpartum
Measure: Number; unit: Percentage of All Household Contacts
Arm/Group | Hospital With Immunization Program | Hospital With No Immunization Program
Number analyzed (Participants) | 238 | 306
Percentage of All Household Contacts | 55 | 39

ADVERSE EVENTS:
Description: Only serious adverse events collected and reported
Arm/Group | Hospital With Immunization Program | Hospital With No Immunization Program
Serious Adverse Events (participants affected / at risk) | 0/238 | 0/306
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No